CLINICAL TRIAL: NCT03579862
Title: Identification and Molecular Characterization of Heritable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: Identification of Heritable CTEPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1024723
Record Dates: First submitted 2018-05-24; First posted 2018-07-09 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
  Interventions: Other: Blood Draw
- Pulmonary Embolism (PE)
  Interventions: Other: Blood Draw
- Pulmonary Arterial Hypertension (PAH)
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw

SUMMARY:
Some patients who have blood clots come down with a life-threatening condition known as Chronic Thromboembolic Pulmonary Hypertension (CTEPH), which is high blood pressure only in the arteries of the lungs. This study seeks to understand more about the genetics causes of CTEPH by obtaining blood samples and examining family histories.

DETAILED DESCRIPTION:
This project proposes to identify a cohort of Utah patients with CTEPH, and to perform a comprehensive analysis of family history and CTEPH risk factors in these patients, and in controls with acute pulmonary embolism (PE) and pulmonary arterial hypertension (PAH). Detailed family history interviews will be performed with all patients, and all enrolled patients will provide a blood sample for thrombophilia testing and for gene sequencing with the goal of identifying novel genetic variants that contribute to CTEPH risk.

ELIGIBILITY:
Inclusion Criteria:

* CTEPH cohort:

  1. Confirmed CTEPH based on having undergone PEA surgery.
  2. Strongly suspected CTEPH based on right heart catheterization data showing mPAP>26 and PCWP<15, and imaging demonstrating chronic thromboembolic disease (either ventilation/perfusion scan, CT pulmonary angiography, or conventional pulmonary angiography).
* PE cohort:

  1. PE diagnosed by CT pulmonary angiography or ventilation/perfusion scan within the preceding 24 months.
  2. No evidence of PH at the time of enrollment (based on absence of dyspnea, exertional chest pain, or exertional presyncope on history, lack of physical exam findings of PH or right heart failure, and lack of signs of PH on objective data including echocardiography and/or right heart catheterization).
  3. No evidence of chronic thromboembolic disease at the time of enrollment (based on chronic appearing thrombus on CT pulmonary angiography or conventional pulmonary angiography, or based on prior high probability ventilation/perfusion scan showing a similar pattern of perfusion defects).
* PAH cohort:

  1. Diagnosis of group 1 PAH.
  2. Prior normal or low probability ventilation/perfusion scan.
  3. No reported history of prior VTE events.
  4. If available, all prior evaluations for VTE (including CT pulmonary angiography and Doppler ultrasound exams) must also be negative.

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CTEPH will be recruited and enrolled at Intermountain Healthcare, also from outside of Intermountain Healthcare, for example at the University of Utah (following IRB approval there) and at national conferences.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2013-12-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of family history of VTE in relatives of CTEPH patients compared to PE and PAH patients in Intermountain populations | through study completion, approximately 18 months

SECONDARY OUTCOMES:
Characteristics of familial and, apparently, sporadic CTEPH in Intermountain populations | through study completion, approximately 18 months
Estimates of prevalence of familial CTEPH in Intermountain populations | through study completion, approximately 18 months
Heritability and penetrance patterns of familial CTEPH | through study completion, approximately 18 months
Discovery and validation of genetic polymorphisms present in familial CTEPH patients | through study completion, approximately 18 months
Identification of gene pathways that may be relevant to the development of CTEPH after actue PE | through study completion, approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dodson, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No